CLINICAL TRIAL: NCT01745640
Title: A Multicenter Open Label Phase II Study of Pomalidomide and Dexamethasone in Progressive Relapsed or Refractory Multiple Myeloma Patients With Deletion 17p or Translocation (4;14) Adverse Karyotypic Abnormalities-IFM2010-02
Brief Title: Pomalidomide and Dexamethasone Effects in Multiple Myeloma Patients With Del 17p or t (4;14)
Acronym: IFM2010-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010_52; 2011-002081-20 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-12-10 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2015-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; dexamethasone; pomalidomide; response; safety; del 17p; t 4-14
MeSH Terms: conditions — Multiple Myeloma; Chromosome 17 deletion | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- POMALIDOMIDE and dexamethasone treatment (Experimental): All patients will receive pomalidomide (4 mg/day per os) and dexamethasone (40/20 mg/wk per os) during 21 day/28 day cycle
  Interventions: Drug: POMALIDOMIDE; Drug: Dexamethasone

INTERVENTIONS:
Drug: POMALIDOMIDE — hard capsule 4mg/day, oral route, from day 1 to 21 per 28 days cycle
  Other Names: 4mg/day, oral route, from day 1 to 21 per 28 days cycle
Drug: Dexamethasone — 40mg (if patient <75 years)/20mg weekly, oral route, on day 1, 8, 15, 22 per 28 days cycle
  Other Names: weekly, oral route, on day 1, 8, 15, 22 per 28 days cycle

SUMMARY:
The purpose of this study is to determine the efficacy and toxicity profile of Pomalidomide and Dexamethasone in relapsed or refractory Multiple Myeloma patients with deletion 17p or translocation (4;14)

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE. Multiple myeloma (MM) is an incurable disease that is characterized by the accumulation of clonal plasma cells in the bone marrow [1]. The median overall survival for patients with myeloma is approximately 4-5 years, and MM remains an incurable disease. Despite front line treatment approaches, the disease eventually relapses. While patients with relapsed disease may achieve responses to subsequent antimyeloma therapies, the duration of response decreases with successive relapses until resistant disease develops. Until recently, the median survival following relapse after induction therapy was approximately one year. The recent US Food and Drug Administration approvals of bortezomib (2003) and combination lenalidomide plus dexamethasone (2006) therapies for the treatment of previously treated MM has provided effective therapeutic options that give patients with relapsed or refractory MM the prospect for a prolongation of overall and progression-free survival times [2-4].

Although the introduction of novel agents to the autologous transplant procedure in patients less than 65 years old or to the Melphalan Prednisone regimen in elderly patients has significantly improved response rates and survival times, MM is a heterogeneous disease with divergent outcomes driven by the biologic characteristics, especially cytogenetic characteristics [5, 6]. Various studies have demonstrated that cytogenetic characteristic as detected by fluorescent in situ hybridization (FISH) was one of the most powerful prognostic marker in MM, especially presence of deletion of 17p13 (del17p) [6, 7] and translocation t(4;14) [6, 7] that represent approximately 20% to 25% of patients in the series [8]. The del(17p) and t(4;14) chromosomal abnormalities are associated with poor progression-free survival and shorter overall survival in newly diagnosed MM patients treated with traditional chemotherapy … The conclusion of recent studies were that a clear unmet medical need still exists for additional novel therapeutic options for the treatment of MM with del17p and t(4;14) and that novel agents should be proposed earlier in the patient evolution.

Pomalidomide belongs to the immunomodulators compounds which thalidomide is the parent compound and lenalidomide the most recently approved agent [14]. It is derived from thalidomide and shares a number of the beneficial pharmacologic properties with thalidomide. The efficacy of thalidomide has been limited by adverse effects, which include sedation, neuropathy, constipation, and deep vein thrombosis. This toxicity profile seems dose and duration-related,which have the potential of improved potency and reduced toxicity. By modifying the thalidomide structure through the addition of an amino group at the 4 position of the phthaloyl ring, pomalidomide was generated.

… A phase 2 randomised open label study of 2 modalities of Pomalidomide plus low-dose Dexamethasone in patients with Multiple Myeloma, refractory to both lenalidomide and bortezomib was conducted. This study was addressed to patients with MM who were symptomatic and progressive following at least two cycles of lenalidomide and two cycles of bortezomib (either separately or in combination). This study provides further evidence that pomalidomide has no-cross resistance with lenalidomide and suggests that it can provide benefit for patients who have relapsed after other novel therapies. This data demonstrated that pomalidomide has significant efficacy in MM and can be safely administered to myeloma patients.

STUDY RATIONALE. There is an increasing number of patients with adverse karyotypic abnormalities, such as del17p and t(4;14), that requires new therapeutic options to improve progression free survival and ultimately overall survival. Based on recent studies, we hypothesized that these patients might benefit from the combination of pomalidomide and dexamethasone. We have therefore designed a Multicenter Open label Phase II study of Pomalidomide and Dexamethasone in Progressive Relapsed or refractory Multiple Myeloma patients with deletion 17p or translocation (4;14) Adverse Karyotypic Abnormalities. This study will determine the efficacy and toxicity profile of pomalidomide and dexamethasone in patients with adverse prognostic factors as determined using adverse karyotypic abnormalities and that are in desperate need of novel therapeutics. This study will be conducted in accordance with "good clinical practice" and all applicable regulatory requirements, including, where applicable, the 2008 version of the Declaration of Helsinki.

STUDY INDICATION In relapsed and refractory MM patients, who are progressive, with MM characterized by Deletion 17p or translocation (4;14) Adverse Karyotypic Abnormalities STUDY DESIGN Overall design. This study is a Multicenter, Open-label, Single arm, Phase 2 study of pomalidomide and dexamethasone in relapsed or refractory MM patients with deletion 17p and translocation (4;14). Eligible patients must have a progressive, relapsed or refractory MM, a deletion 17p and/or translocation (4;14) using FISH technique and a measurable disease. There is no escalation dose study, the Maximum Tolerated Dose has already been determined in previous phase 1-2 escalation dose studies as 4 mg/day on day 1 to 21 of a 28 days cycle. The proposed dose of dexamethasone is considered standard. Patients will receive the pomalidomide and dexamethasone regimen until progression. This study will eventually improve time to disease progression and response rates, with no additional toxicity, as compared to other available regimens, in this subgroup of patients with myeloma characterized with an adverse prognosis.

Regimen Pomalidomide 4mg/day, oral route, from day 1 to 21 per 28 days cycle Dexamethasone 40mg weekly, oral route, on day 1, 8, 15, 22 per 28 days cycle for patients aged less than 75 years, and 20 mg once weekly oral route per 28 days cycle for patients aged 75 years and above.

Until progression either relapse or refractory.

Potentially eligible patients and informed of their rights and how to achieve the study will sign informed consent prior to undergoing any study-related procedures. Patients will undergo screening assessments for protocol eligibility within 28 days of randomization.

For all patients who enroll into this study, study visits and serial measurements of safety and efficacy will be performed on a monthly basis for the first 12 months then on a 2-months basis thereafter. Tumor response, including progressive Disease, will be assessed according to the IMWG criteria. The severity of Adverse Events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0. In this study, a central laboratory will analyze serum and urine protein electrophoresis tests (myeloma [M]-protein levels), serum and urine immunofixation studies (CHRU Lille). FISH cytogenetic will be performed in Nantes for all patients in the study.

Efficacy assessments will occur on a monthly basis (28 days, designated as Study Day) for the first 12 months then on a 2-months basis thereafter, regardless of current cycle day, and can be performed within 3 days to day one of the cycle. Study of vital signs and performance status is requested at Study Day.

Study Day 1 of Open-Label Treatment will occur on the day the patient starts the pomalidomide-dexamethasone regimen. This regimen is given on oral route for the 2 therapeutic agents tested. complete blood (cell) count will be monitored at least every 7 days (weekly) during the first cycle. It will also be monitored at the first day of each cycle thereafter.

Recommended concomitant therapy. All medications (prescription and non-prescription), treatments and therapies taken from 28 days prior to initiation of the study through the last dose of study drug, must be recorded in the case report form. Any treatments or therapies used to treat a Serious Adverse Event that occur within 28 days of discontinuation of study drug must also be documented.

In addition, all patients will be given prophylactic anti-thrombotic treatment, either aspirin daily (commercial supply) if the patient has no prior history of thrombosis events or low molecular weight heparin according to hospital guidelines or physician preference. All prophylactic antithrombotic treatment unless contraindicated according to hospital guidelines or physician preference must be recorded. All patients will be monitored for signs and symptoms of venous thromboembolism while on Pomalidomide.

The use of hematopoietic growth factors is permitted during the study. The use of bisphosphonates is permitted throughout the study at the discretion of the Investigator.

Other therapies considered necessary for the patient's well being may be administered at the discretion of the Investigator. These therapies may include antibiotics, analgesics, antihistamines, or other medications and transfusions of red blood cells, platelets, or fresh frozen plasma given to assist in the management of complications associated with multiple myeloma or its therapy.

Prohibited concomitant therapy Concomitant use of sargramostim, other anti-cancer therapies, including thalidomide, or other investigational agents is not permitted while subjects are receiving study drug of the study. The need for radiation therapy is considered to be a treatment failure. However, an exception (that is patients allowed to remain in the treatment phase of the study) is made for radiation therapy to a pathological fracture site to enhance bone healing or to treat post-fracture pain that is refractory to narcotic analgesics because pathologic bone fractures do not by themselves fulfill a criterion for disease progression End of study treatment. Patients may continue study treatment until Progression develops (last study drug intake of pomalidomide-dexamethasone regimen) at which time they will complete a Treatment Discontinuation visit as outlined in Table 2.

Follow-Up. Upon discontinuation from pomalidomide-dexamethasone study treatment for Progression or any other reason, patients will be assessed for 28 days. Serious Adverse Events will continue to be collected on patients during the first 28 days in Follow-Up. FCBP will have a final pregnancy test 28 days after the last dose of study drug if they have regular or no menstrual cycles; or 14 and 28 days after the last dose if menstrual cycles are irregular. In addition, patients who are discontinued from study treatment will be followed for overall survival and subsequent MM treatment regimens.

Patients who discontinue treatment for other reason than Progression will have response determined until Progression or until start of further myeloma therapy.

All patients will have survival data entered in the Case Report Form after progression, along with subsequent myeloma treatments.

Dose Interruption and Modification. Dose interruption and reduction for pomalidomide-dexamethasone regimen will be provided.

PHASE OF DEVELOPMENT 2 STUDY PRODUCTS This is a single arm phase 2 study. Each patient will receive 28 day cycles of Pomalidomide and Dexamethasone treatment until progression, either relapse or refractory.

Pomalidomide 4mg/day, oral route, from day 1 to 21 per 28 days cycle Dexamethasone 40mg weekly, oral route, on day 1, 8, 15, 22 per 28 days cycle for patients aged less than 75 years, and 20 mg once weekly oral route per 28 days cycle for patients aged 75 years and above.

Dose adaptation will be provided within the protocol

ELIGIBILITY:
inclusion criteria:

* Able to understand and voluntarily sign an informed consent form
* Age >18 years
* Life expectancy > 6 months.
* Patients must have a Symptomatic and Progressive MM
* Patients must have a clearly detectable and quantifiable monoclonal M-component value
* Eastern Cooperative Oncology Group performance status score of 0, 1, or 2
* Adequate bone marrow function, with no transfusion within 5 days prior to treatment.
* Adequate organ function
* Wash out period of at least 2 weeks from previous antitumor therapy or any investigational treatment.
* Able to take antithrombotic medicines
* Subjects affiliated with an appropriate social security system.
* Agree to abstain from donating blood while taking study drug therapy and for at least 28 days following discontinuation of study drug .
* Female subjects of childbearing potential (FCBP) (*) must:

Understand the potential teratogenic risk of the treatment and take the relative precaution mentioned in the protocol, in the Pomalidomide information sheet Agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation

* For female NOT of childbearing potential, pomalidomide is contraindicated unless the exceptions mentioned in the protocol
* Understand the hazards and necessary precautions associated with the use of pomalidomide
* Male subjects must:
* Understand the potential teratogenic risk and take the relative precaution mentioned in the protocol, in the Pomalidomide information sheet

Exclusion criteria :

* Patient that will require allogeneic or autologous transplantation following pomalidomide dexamethasone treatment while in the same course.
* Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation
* Use of any other experimental drug or therapy within 15 days of screening.
* Patients with renal failure that require dialysis and patients with creatinine clearance < 50 mL/min
* Prior history of malignancies, other than multiple myeloma, unless the patients has been free of the disease for ≥3 years. Excepted those mentioned in the protocol.
* Prior local irradiation within two weeks before screening
* Ongoing active infection, especially ongoing pneumonitis
* Ongoing Cardiac dysfunction
* Inability or unwillingness to comply with birth control requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (from the date of the first dose to the date of the first observation of disease progression) | The final analysis of disease progression will be run when at least 29 events will occur (expected average of 32months ).
  The time to progression (TTP) is the time from the start of treatment to the first documentation of disease progression or death from any cause during study, whichever occurs earlier.The Kaplan-Meier procedures will be used to characterize the time-to-event curves (TTP, OS, response duration and EFS) when there is censoring; univariate summary statistics will be provided for time to response.

SECONDARY OUTCOMES:
Safety of pomalidomide and dexamethasone | for the first 15 patients included at time they end cycle 1 (an expected average of 6 months from the first inclusion)
  All patients who receive at least one dose of study medication will be included in the safety analyses. Adverse events, vital sign measurements, clinical laboratory information, and concomitant medications will be tabulated and summarized when appropriate.
  Patient incidence rates of all Adverse Events will be tabulated by body system class, preferred term, and severity grades whenever possible and will be provided with the number and percentage of subjects with adverse events
Overall Response rate (Partial Response and better), Very Good Partial Response (VGPR) + Complete Response (CR) rate and stringent Complete Response (sCR) rate to pomalidomide and dexamethasone in MM patients | The final analysis of disease progression will be run when at least 29 events will occur (expected average of 32months from beginning of study ).
  Response rate (Partial Response and better) to pomalidomide and Dexamethasone in the studied population will be determined using International Myeloma Working Group (IMWG) response criteria. VGPR + CR rate and sCR rate will also be determined using IMWG [1]
Time to response and Response duration of pomalidomide and dexamethasone. | The final analysis of disease progression will be run when at least 29 events will occur (expected average of 32months from beginning of study ).
  A responder will be any patient who shows at least a partial response (PR) at any time during the study. For responders, time to response and response duration will be analyzed. Time to response is the time from the start of treatment to the first documentation of response (either PR or better). Duration of response is the time from the first PR or better to the first documentation of disease progression. Following the completion of the first cycle, efficacy assessments will be given every 28 days as long as they stay on treatment up to 12 months then every 2 months until progression.
Overall Survival of pomalidomide and dexamethasone and event free survival | The final analysis of disease progression will be run when at least 29 events will occur (expected average of 32months from beginning of study ).
  The median overall survival for patients with MM is approximately 4-5 years, and MM remains an incurable disease. Overall survival (OS) is the time from the start of treatment to date of last news or death from any cause. Event free survival (EFS) is the time from the start of treatment to the date of progression, death, or other cause of discontinuation of study drug, including serious drug toxicity.
Response and Time to disease progression with regards to cytogenetic abnormalities in the bone marrow tumor plasma cells | The final analysis of disease progression will be run when at least 29 events will occur (expected average of 32months from beginning of study ).
  Response rate (Partial Response and better) to pomalidomide and Dexamethasone in the studied population will be determined using International Myeloma Working Group (IMWG) response criteria. VGPR + CR rate and sCR rate will also be determined using IMWG [1]

CONTACTS AND LOCATIONS:
Overall Officials: Xavier LELEU, PHD, Principal Investigator — CHRU de Lille
Locations (20):
- France (20):
  - CHRU-Hôpital Sud Amiens, Amiens
  - Chru Caen, Caen
  - CHU DIJON, Hôpital d'Enfants, Dijon
  - CHRU, Hôpital A.Michallon, Grenoble
  - Centre hospitalier départemental La Roche sur Yon, La Roche-sur-Yon
  - Chru Lille, Lille
  - Institut Paoli Calmette,, Marseille
  - CHRU, Hôtel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU - Hôpital St Antoine,, Paris
  - Hôpital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud -1, Pierre-Bénite
  - Centre Hospitalier Lyon Sud -2, Pierre-Bénite
  - CHRU POITIERS-Hôpital Jean Bernard, Poitiers
  - Hôpital Robert Debré, CHU Reims, Reims
  - CHRU RENNES 2, Hôpital Pontchaillou, Rennes
  - CHRU RENNES 1, Hôpital Sud, Rennes
  - CHRU, Hôpital Purpan, Toulouse
  - CHRU- Hôpital Bretonneau, Tours
  - CHRU, Hôpitaux de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Leleu X, Karlin L, Macro M, Hulin C, Garderet L, Roussel M, Arnulf B, Pegourie B, Kolb B, Stoppa AM, Brechiniac S, Marit G, Thielemans B, Onraed B, Mathiot C, Banos A, Lacotte L, Tiab M, Dib M, Fuzibet JG, Petillon MO, Rodon P, Wetterwald M, Royer B, Legros L, Benboubker L, Decaux O, Escoffre-Barbe M, Caillot D, Fermand JP, Moreau P, Attal M, Avet-Loiseau H, Facon T; Intergroupe Francophone du Myelome (IFM). Pomalidomide plus low-dose dexamethasone in multiple myeloma with deletion 17p and/or translocation (4;14): IFM 2010-02 trial results. Blood. 2015 Feb 26;125(9):1411-7. doi: 10.1182/blood-2014-11-612069. Epub 2015 Jan 9. PMID 25575538